CLINICAL TRIAL: NCT03468647
Title: FRAGIL-IT, Seamless Follow up and Support System for Frail Elderly Living at Home
Brief Title: Seamless Follow up and Support System for Frail Elderly Living at Home
Acronym: FRAGIL-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC31/15/0603
Record Dates: First submitted 2017-10-13; First posted 2018-03-16 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Elderly
Keywords: frailty; tele-monitoring; self-management
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FRAGIL-IT testing group (Experimental): FRAGIL-IT tools : connected soles, connected weighting machine and measure of gripping force
  Interventions: Other: soles; Other: weighting machine; Other: gripping force

INTERVENTIONS:
Other: soles — Volunteer must walk this this connected seamless to measure different walking parameters
  Other Names: connected soles
Other: weighting machine — This weighting machine measure weight evolution and equilibrate of volunteers
  Other Names: connected weighting machine
Other: gripping force — this machine measure the gripping force of volunteer
  Other Names: gripping force machine

SUMMARY:
The object of the present project is to promote the prevention of disability by providing 1) a feedback and motivational coaching to the user, 2) relevant clinical parameters to the healthcare professionals in order to support the patient's follow-up, and 3) supporting the detection of preliminary signs of functional loss. The technical solution will contain wearable (e.g. smart insole) and ambient unobtrusive devices (e.g. weigh scale including balance analysis), and analysis and diagnosis assistance software. The devices transmit wirelessly the collected data to a remote server through a tablet. Data will then be available remotely for consultations by users (i.e. patients or physicians). The clinical evaluation will be a multi-phased design with a first living lab evaluation followed by a real life home trial to finalize the evaluation. Comprehensive assessments will be conducted to highlight the feasibility and acceptability.

DETAILED DESCRIPTION:
Functional decline challenges the sustainability of healthcare systems. There are difficulties in implementing effective interventions to prevent disability, to promote adherence to lifestyle recommendations and to perform seamless follow-up at home. A technological solution addressing this challenge and improving individual participation would be welcome. Our aim is to evaluate an instrument for supporting physical activity and monitoring multiple parameters of frailty (a pre-disability condition) in frail elderly persons. The investigator and collaborator are therefore developing a solution to monitor key parameters of frailty during subject daily life and to promote walking. This tools are :

1. connected soles to evaluate different parameters of the volunteer walking
2. connected weighing machine to evaluate the volunteer weight and equilibrate
3. machine to measure gripping force because gripping force is correlated to physical condition.

The primary aim is to assess the acceptability of the solution for the follow up and the motivational coaching of frail patients at home. Results from this study will also be used to elaborate the design of a further larger national multicenter randomized control trial assessing the efficiency of the solution to prevent disability.

ELIGIBILITY:
Inclusion Criteria:

* patient living at home;
* pre-frail or frail volunteers;
* Informed and written consent by the patient or the legal representative or the reliable person when appropriate.

Exclusion Criteria:

* patient's life expectancy less than 12 months; patient presenting disability with an Activity of Daily Living score < 4/6 ant/or a Mini - Mental State <20/30, not walking or walking with a technical support;
* Non agreement of study participation of patients or legal representative or the reliable person when appropriate.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
acceptability of FRAGIL-IT tools | 3 months
  primary outcome is based on the acceptability of the FRAGIL-IT tools for the end-user : connected soles, connected weighting machine and measure of gripping force to control autonomy loss. The acceptability of this tools will be evaluate by questionnaire as The Short Form (36) Health Survey (SF36) questionnaire

SECONDARY OUTCOMES:
evaluation of life quality with SF36 questionnaire | 3 months
  the life quality will be assess with SF36 questionnaire
functional status measure by ADL | 3 months
  functional status will be assess with Activity of Daily Living (ADL) score. The scale of ADL is between 0 to 6. 0 is worse than 6.
functional status measure by iADL | 3 months
  functional status will be assess with instrumental Activity of Daily Living (iADL) score. The scale of IADL is between 0 to 8. 0 is worse than 8.
cognitive status | 3 months
  cognitive status will be assess with Mini Mental State (MMS)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine PIAU, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital, Toulouse, Toulouse, Midi-Pyrenes, France